CLINICAL TRIAL: NCT01803750
Title: Building a Network of Community Primary Care Providers to Implement and Disseminate Cancer Prevention Interventions for Latino Populations
Brief Title: Community Primary Care Providers to Implement and Disseminate Cancer Prevention Interventions for Latino Populations
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13-031
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: For New York State Registered Family Practitioners and Internal Medicine Physicians
Keywords: Primary Care Providers; Latino Populations; Disseminate Cancer Prevention; semi-structured interviews; 13-031

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Primary Care Providers: Conduct and analyze in-depth, semi-structured interviews with community-based primary care providers serving large Latino populations and Form a community-based participatory committee.
  Interventions: Behavioral: in-depth, semi-structured interviews

INTERVENTIONS:
Behavioral: in-depth, semi-structured interviews — In-depth interviews will be conducted by the Principle Investigator and will use a combination of open-ended and closed, fixed response questions. Interviews will be audio recorded if the participant agrees, and answers to fixed response questions will be marked for complete analysis. The data collection portion of the study is estimated to take approximately 8 months. Areas to be addressed in the open-ended portion of the interview include: 1) Knowledge, attitudes and beliefs toward evidence-based cancer screening and prevention approaches 2) Barriers to implementing evidence-based cancer screening practices in the individual provider's clinical setting 3) Preferences for mechanisms of information dissemination and implementation and 4) Ideas and methods to facilitate evidence-based practices to improve cancer screening in the Latino population. A community-based participatory committee (CBPC) will be formed with 5-7 key informants identified during the interview process.

SUMMARY:
The purpose of this study is to understand primary care provider's knowledge, attitudes, and barriers to promoting evidence-based cancer screening and prevention practices for physicians with large Latino patient populations. The investigators will ask providers information on cancer screening and prevention practices by conducting one-on-one interviews. In addition, they would like to develop a committee of community providers to help design and implement cancer screening and prevention programs specifically for Latino patients based on the interview findings.

ELIGIBILITY:
Inclusion Criteria:

* New York State registered family practitioners and internal medicine physicians
* Minimum one half of their patients are Latino (provider self-reported)
* Currently practice in a small clinical setting (defined by no more than 5 providers) including community clinics, and/or private practice in Queens, Brooklyn, Bron and Staten Island, New York
* No active affiliation with a major hospital or academic institution.

Exclusion Criteria:

* Practicing medicine for less than 2 years
* Practicing in a setting where no health insurance is accepted

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be primary care providers (PCPs) in the NYC Queens. Brooklyn ,Bronx and Staten Island, borough neighborhoods that serve large Latino populations.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
assess attitudes and barriers | 1 year
  of community-based primary care providers serving large Latino patient populations toward implementing evidence-based practices for cancer screening and prevention.

SECONDARY OUTCOMES:
build the beginning of a Community-Based Participatory Committee | 1 year
  and determine the feasibility of a network of community primary care providers serving large Latino patient populations with the purpose of disseminating, implementing and evaluating evidence-based practice for cancer screening and prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Aragones, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/